CLINICAL TRIAL: NCT07200414
Title: Strengthening HPV Vaccination and Adolescent Health Research Program in Nigeria (SHARP in Nigeria)
Brief Title: Strengthening HPV Vaccination and Adolescent Health Research Program in Nigeria (SHARP)
Acronym: SHARP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Direct Consulting and Logistics (Unknown); Jhpiego (Other); Gavi, The Vaccine Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00030748
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Human Papillomavirus (HPV) Vaccine; Human Papillomavirus (HPV) Vaccines; Human Papillomavirus (HPV) Infections; Adolescent Health Services
Keywords: HPV vaccination uptake; Nigeria; Human Papillomavirus; Vaccination coverage; Adolescents; Adolescent Health Services; Immunization programs; Health Services Accessibility
MeSH Terms: conditions — Papillomavirus Infections; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Adolescent Health Package (Experimental): Local government areas (LGAs) where the routine government health system delivers an integrated package of adolescent health services. The package includes HPV vaccination, sexual and reproductive health counseling, general health check-ups, nutrition and vision screening, mental health support, deworming, and dental and oral health services.
  Interventions: Behavioral: Integrated Adolescent Health Package
- Standard Services (Active Comparator): Local government areas (LGAs) where only standard government health services are provided. HPV vaccination and other adolescent health services are delivered according to routine practice without the additional integrated package.
  Interventions: Other: Routine Government Health Services

INTERVENTIONS:
Behavioral: Integrated Adolescent Health Package — Delivery of an integrated package of adolescent health services through government health facilities. The package includes HPV vaccination, sexual and reproductive health counseling, general health check-ups, nutrition and vision screening, mental health support, deworming, and dental and oral health services. Implemented in intervention LGAs in Lagos and Kebbi States.
  Other Names: SHARP Integrated Package; Integrated Package of Adolescent Services
  Arms: Integrated Adolescent Health Package
Other: Routine Government Health Services — Routine government health services provided in comparison LGAs. Services may include HPV vaccination as per national immunization schedules and other adolescent health services delivered under existing programs, but without the integrated package.
  Other Names: Standard Services
  Arms: Standard Services

SUMMARY:
The goal of this clinical trial is to learn whether adding adolescent health services to routine government health programs can increase Human Papillomavirus (HPV) vaccination coverage among 9-year-old girls and improve use of other health services by adolescents in Nigeria. The main questions it aims to answer are:

Does offering an integrated package of adolescent health services increase the proportion of 9-year-old girls who receive the HPV vaccine?

Does this package increase use of other services such as reproductive health counseling, nutrition and vision screening, mental health services, and deworming among girls and boys ages 9-15 years?

Researchers will compare areas that receive the integrated package to areas that continue with the standard government services to see if the intervention improves vaccination and health service use.

Participants will:

Be surveyed about HPV vaccination and health service use before and after the program is offered.

Take part in interviews or focus groups about experiences with adolescent health services.

Be offered HPV vaccination and other adolescent health services through local health facilities.

DETAILED DESCRIPTION:
This is a mixed-methods, quasi-experimental implementation science study to evaluate the integration of adolescent health services with routine HPV vaccination in Nigeria. The study is being conducted in Lagos and Kebbi States between October 2024 and December 2025.

The intervention will leverage the routine government health system to deliver an integrated package of adolescent health services that includes HPV vaccination and additional services such as sexual and reproductive health counseling, general health check-ups, nutrition and vision screening, mental health services, deworming, and dental and oral health care.

The primary objective is to determine the effect of the integrated package on HPV vaccine coverage among 9-year-old girls. Secondary objectives include: (1) assessing changes in uptake of other adolescent health services among girls and boys aged 9-15 years, (2) examining feasibility, acceptability, and fidelity of the intervention from the perspective of adolescents, parents, providers, and policymakers, and (3) estimating incremental costs of delivering the integrated package.

The study design includes three phases: formative research, implementation, and evaluation. Baseline and endline household surveys will be conducted with parents and adolescents, supplemented by qualitative data collection (in-depth interviews (IDI), focus groups, key informant interviews (KII), and multi-informant interviews (MII)). Service delivery records and costing data from 30 health facilities will also be analyzed.

Comparison will be made between intervention and comparison local government areas to assess differences in HPV vaccine uptake and adolescent health service utilization. The study will generate evidence on strategies to improve HPV vaccination coverage and strengthen adolescent health service delivery in Nigeria.

ELIGIBILITY:
Inclusion Criteria:

* Immunization program managers from National Primary Health Care Development Agency of Nigeria (NPHCDA), state and Local Government Area (LGA) must:
* Have at least one year of experience in current position
* Be part of the HPV vaccine working group and be engaged in discussions around the HPV routinization plan.
* Be involved in the Routine Immunization (RI) working group at the national or state level, or be part of the local government (LG) RI team, and participate in regular discussions about the HPV vaccination program
* Have been involved in the HPV vaccine rollout, including planning, training, deployment, fieldwork, or assessment activities.
* Must be knowledgeable about vaccination programs in the country and able to provide valuable insights into service delivery practices at different levels.

Program managers from the Ministries of Health, and Education must:

* Have at least one year of experience in current position
* Be knowledgeable about adolescent health programs or policies as it relates to the Ministry and its engagements with Ministry of Health and NPHCDA

Health service providers must:

* Have at least one year of experience in current position
* Provide immunization services at the facility, school or community levels
* Have been involved in the HPV vaccine rollout, including planning, training, deployment, fieldwork, or assessment activities.
* Must be knowledgeable about vaccination programs in the country and able to provide valuable insights into service delivery practices at different levels.

School-based service providers such as principals, teachers and school nurses must:

* Have at least one year of experience in current or similar roles within the educational system.
* Have previous involvement or interest in school health initiatives, adolescent health issues, including sexual health education, vaccination programs etc.
* Be employed in schools located within Lagos or Kebbi states where adolescent girls (9-15 years) attend
* Be a representative from public, private, urban or rural schools, including those serving underprivileged students.
* Be willing to participate in interviews and share experiences and opinions.
* Be proficient in English or Yoruba for Lagos, or English or Hausa for Kebbi

Civil Society Organization (CSO) partner in the state must:

* Be engaged in any of the following cervical cancer elimination, HPV vaccination, girl-child education, internally displaced persons rehabilitation, and youth empowerment within the last 2 years in the intervention LGAs
* Have working relationship with the immunization program at the national, state, local or ward level

Adolescent male and female respondents:

* Must be aged between 9-19 years for the HCD workshop, (In-Depth Interview) IDIs and FGDs, and aged between 9-15 years for the household surveys
* Must reside in the study states (Lagos or Kebbi and in the study LGAs) to be considered for all data collection activities,
* Must have parental or guardian consent to participate in all data collection activities unless classified as emancipated minors.
* In addition to having parental or guardian consent, adolescents must be willing to participate in the data collection activities.
* Adolescents aged 9 to 17, who are legally considered emancipated (e.g. married) can provide consent for participation in all data collection activities without requiring parental or guardian consent
* Must not have participated in any other data collection activity in the study, since distinct adolescents will be enrolled for each data collection activity.

Parents must:

* Be parents or legal guardians of adolescents aged 9-19 years.
* Reside in Lagos or Kebbi states.
* Be willing to participate in the interview process and share experiences, concerns, and suggestions.
* Be proficient in English or Yoruba for Lagos, or English or Hausa for Kebbi.

Community leaders:

* Have at least one year of experience in current role
* Reside in Lagos or Kebbi states
* Must be residing in the community for more than 1 year
* Be willing to participate in the interview process and share experiences, concerns, and suggestions.
* Be proficient in English or Yoruba for Lagos, or English or Hausa for Kebbi.

Exclusion Criteria:

1. For all participants

   * Individuals unable to participate due to time constraints or conflicting responsibilities.
   * Those not proficient in the necessary languages (English or Yoruba for Lagos, English or Hausa for Kebbi).
   * For the Key Informant Interviews (KIIs), Multi-Informant Interviews (MIIs), Focus Group Discussions (FGDs) and Household Surveys (HHS): sub-national level individuals not residing in the respective study states (Lagos and Kebbi)
   * For the Human-Centered Design Workshop (HCD) workshop: LGA, ward, facility, community, school-level participants who are not from the intervention LGA
   * Those who do not provide consent or assent.
   * Those who lack the capacity to provide consent or assent or participate effectively
2. For specific participant types

   * Immunization program managers from NPHCDA, state and LGA levels
   * Individuals with less than one year experience in current position and in immunization programs.
   * Those who have not been involved in HPV vaccination program operations or lack a comprehensive view of potential service delivery options.
   * Program managers who do not belong to the National or state or LGA or Ward HPV Technical Working Group
   * Program managers from the Ministry of Health, Women affairs and Education
   * Individuals with less than one year experience in current position.

Health service providers:

* Healthcare workers who didn't participate in the HPV vaccine introduction and has less than 1 year working in routine immunization.
* School-based service providers such as principals, teachers and school nurses
* Individuals without experience teaching adolescents 9-15 years or lacking familiarity with the educational system.
* Teachers or principals from institutions not relevant to the study, such as boys-only school, or universities.

Adolescents:

* Adolescents outside the specified age range of 9-19 years.
* Those unable to communicate effectively, even with interpreters or accommodation.
* Adolescents with medical conditions preventing participation in discussions about vaccination or health.
* Those whose parents or guardians do not provide consent or who do not assent to participate.
* Wards of the state or adolescent under government supervision

Parents:

* Individuals who are not parents or guardians of adolescents aged 9-15 years.
* Parents with extreme beliefs or conspiracy theories about vaccinations that may not contribute constructively to the program design process (For HCD only)
* School teachers in only boys' school or girls outside the age range of 9-15 years.
* Community influencers that have resided in the community for less than one year

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14768 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in HPV vaccine coverage among 9-year-old girls from baseline to endline | Baseline, 14 months
  Human Papillomavirus Virus (HPV) vaccine coverage will be assessed among 9-year-old girls in intervention and comparison (Local Government Areas (LGAs) using baseline and endline household surveys of mother-daughter dyads, supported by administrative vaccination records from health facilities. Differences between baseline and endline coverage in intervention LGAs will be compared with those in comparison LGAs to estimate the impact of the integrated adolescent health package.
Proportion of 9-year-old girls who received at least one dose of HPV vaccine | Baseline, 14 months
  Assessed using baseline and endline household surveys and service delivery data. Coverage will be calculated as the number of eligible girls who received at least one dose divided by the total eligible girls surveyed.

SECONDARY OUTCOMES:
Proportion of adolescents aged 9-15 who report use of at least one adolescent health service | Baseline, 14 months
  Services may include Sexual and Reproductive Health (SRH) counseling, nutrition or vision screening, mental health services, deworming, or dental/oral care. Measured using baseline and endline household surveys and service records.

CONTACTS AND LOCATIONS:
Overall Officials: Chizoba Wonodi, MBBS, DrPH, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Lagos State Ministry of Health/Kebbi State Ministry of Health, Lagos, Nigeria

REFERENCES:
- [Background] Adeyanju GC, Essoh TA, Sidibe AR, Kyesi F, Aina M. Human Papillomavirus Vaccination Acceleration and Introduction in Sub-Saharan Africa: A Multi-Country Cohort Analysis. Vaccines (Basel). 2024 May 1;12(5):489. doi: 10.3390/vaccines12050489. PMID 38793741
- [Background] Lawson O, Ameyan L, Tukur Z, Dunu S, Kerry M, Okuyemi OO, Yusuf Z, Fasawe O, Wiwa O, Hebert KS, Joseph JT, Nwokwu UE, Okpako O, Chime CI. Cervical cancer screening outcomes in public health facilities in three states in Nigeria. BMC Public Health. 2023 Sep 1;23(1):1688. doi: 10.1186/s12889-023-16539-1. PMID 37658293
- [Background] Singh D, Vignat J, Lorenzoni V, Eslahi M, Ginsburg O, Lauby-Secretan B, Arbyn M, Basu P, Bray F, Vaccarella S. Global estimates of incidence and mortality of cervical cancer in 2020: a baseline analysis of the WHO Global Cervical Cancer Elimination Initiative. Lancet Glob Health. 2023 Feb;11(2):e197-e206. doi: 10.1016/S2214-109X(22)00501-0. Epub 2022 Dec 14. PMID 36528031